CLINICAL TRIAL: NCT02393352
Title: Benefits of Dry Needling in Trigger Points on Autonomic Nervous System, Photoelectric Plethysmography, Body Composition in Patients With Fibromyalgia Syndrome.
Brief Title: Benefits of Dry Needling in Trigger Points on Autonomic Nervous System and Corporal Composition in Patients With Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD (Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UAL_435
Record Dates: First submitted 2015-03-04; First posted 2015-03-19 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Fibromyalgia; Trigger Points
Keywords: Body Composition; Autonomic Nervous System; Oxygen; Randomized Controlled Trial
MeSH Terms: conditions — Fibromyalgia | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Needling Therapy (Experimental): The dry needling therapy will be applied on active trigger points in occipital muscle, splenius capitis, sternocleidomastoid muscle, scalene muscles, trapezius, supraspinatus, infraspinatus muscle, latissimus dorsi, iliocostalis muscle, multifidus muscles, and quadratus lumbourm muscles.
  Interventions: Other: Dry Needling Therapy
- Electrical Stimulation Therapy (Active Comparator): Diadynamic fixed current phase in active trigger points, with pulses of 10msec, and intervals of equal duration.
  Interventions: Other: Electrical Stimulation Therapy

INTERVENTIONS:
Other: Dry Needling Therapy — The dry needling therapy will be applied on active trigger points in occipital muscle, splenius capitis, sternocleidomastoid muscle, scalene muscles, trapezius, supraspinatus, infraspinatus muscle, latissimus dorsi, iliocostalis muscle, multifidus muscles, and quadratus lumbourm muscles.
  Arms: Dry Needling Therapy
Other: Electrical Stimulation Therapy
  Arms: Electrical Stimulation Therapy

SUMMARY:
This study evaluates the benefits of dry needling in trigger points on autonomic nervous system, photoelectric plethysmography, body composition in patients with fibromyalgia syndrome.

DETAILED DESCRIPTION:
Dru needling can be developed on active trigger points. Myofascial trigger points can be active or latent. An active myofascial trigger point pain causes giving a specific pathological picture. We will conduct a location of myofascial trigger points following the illustrations location myofascial trigger points that indicate Travell and Simons both left-sided and right.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia syndrome diagnosis.
* Aged from 18 to 65 years.
* No regular physical activity.
* Limitation of usual activities due to pain on at least 1 day in the previous 30 days.
* Agreement to attend evening therapy sessions.

Exclusion Criteria:

* Severe physical disability.
* Comorbid conditions (eg, morbid obesity, inflammatory diseases, irritable bowel syndrome, interstitial cystitis).
* Uncontrolled endocrine disorders (eg, hyperthyroidism or hypothyroidism, diabetes).
* Malignancy.
* Psychiatric.
* Illnesses (eg, schizophrenia or substance abuse).
* Medication usage other than as-needed analgesics (excluding long-term narcotics).
* History of surgery.
* History of whiplash injury.
* Presence of a score >9 points in the Beck Depression Inventory.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Changes Scores on Visual Analoge Scale | At baseline and 4 weeks
  Intensity of pain (within McGill questionnaire)

SECONDARY OUTCOMES:
Changes Scores on Percentage Evaluation Peripheral Capillary Oxygen saturation and photoelectric plethysmograph (Analysis of pulse wave and PANI) | At baseline and 4 weeks
  Cardiac output. Reflectivity index. Stiffness index. Oxygen saturation.
Change Scores on Body Composition | At baseline and 4 weeks
  Fat mass. Body fat mass. Intracellular water. Extracellular water. Fat-free mass. Total body water.
Changes Scores on Cholinergic response indicators (%). | At baseline and 4 weeks
Changes Scores on Heart rate variability. | At baseline and 4 weeks
Changes Scores on Valsalva ratio. K30/15. | At baseline and 4 weeks
Changes Scores on Systemic vascular resistance. | At baseline and 4 weeks
Changes Scores on Systolic pressure. | At baseline and 4 weeks
Changes Scores on Diastolic pressure. | At baseline and 4 weeks
Changes Scores on Assessment of autonomic nervous system | At baseline and 4 weeks
  Galvanic response estimate.

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaida María Castro-Sánchez, Almería, Spain

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Arnold LM, Clauw DJ, McCarberg BH; FibroCollaborative. Improving the recognition and diagnosis of fibromyalgia. Mayo Clin Proc. 2011 May;86(5):457-64. doi: 10.4065/mcp.2010.0738. PMID 21531887
- [Background] Goldenberg DL. Fibromyalgia syndrome: an emerging but controversial condition. JAMA. 2014 Apr 16;311(15):1570. doi: 10.1001/jama.2013.279453. No abstract available. PMID 24737378
- [Background] Castro-Sanchez AM, Mataran-Penarrocha GA, Sanchez-Labraca N, Quesada-Rubio JM, Granero-Molina J, Moreno-Lorenzo C. A randomized controlled trial investigating the effects of craniosacral therapy on pain and heart rate variability in fibromyalgia patients. Clin Rehabil. 2011 Jan;25(1):25-35. doi: 10.1177/0269215510375909. Epub 2010 Aug 11. PMID 20702514
- [Background] Hidalgo-Lozano A, Fernandez-de-las-Penas C, Diaz-Rodriguez L, Gonzalez-Iglesias J, Palacios-Cena D, Arroyo-Morales M. Changes in pain and pressure pain sensitivity after manual treatment of active trigger points in patients with unilateral shoulder impingement: a case series. J Bodyw Mov Ther. 2011 Oct;15(4):399-404. doi: 10.1016/j.jbmt.2010.12.003. Epub 2011 Jan 17. PMID 21943613
- [Background] Pastor Mira MA, Lledo Boyer A, Lopez-Roig S, Pons Calatayud N, Martin-Aragon Gelabert M. [Predictors of healthcare resource use in fibromyalgia]. Psicothema. 2010 Nov;22(4):549-55. Spanish. PMID 21044477
- [Background] Castro-Sanchez AM, Mataran-Penarrocha GA, Granero-Molina J, Aguilera-Manrique G, Quesada-Rubio JM, Moreno-Lorenzo C. Benefits of massage-myofascial release therapy on pain, anxiety, quality of sleep, depression, and quality of life in patients with fibromyalgia. Evid Based Complement Alternat Med. 2011;2011:561753. doi: 10.1155/2011/561753. Epub 2010 Dec 28. PMID 21234327
- [Background] Giamberardino MA, Affaitati G, Fabrizio A, Costantini R. Effects of treatment of myofascial trigger points on the pain of fibromyalgia. Curr Pain Headache Rep. 2011 Oct;15(5):393-9. doi: 10.1007/s11916-011-0205-3. PMID 21541831
- [Background] Affaitati G, Costantini R, Fabrizio A, Lapenna D, Tafuri E, Giamberardino MA. Effects of treatment of peripheral pain generators in fibromyalgia patients. Eur J Pain. 2011 Jan;15(1):61-9. doi: 10.1016/j.ejpain.2010.09.002. PMID 20889359
- [Background] Alonso-Blanco C, Fernandez-de-Las-Penas C, de-la-Llave-Rincon AI, Zarco-Moreno P, Galan-Del-Rio F, Svensson P. Characteristics of referred muscle pain to the head from active trigger points in women with myofascial temporomandibular pain and fibromyalgia syndrome. J Headache Pain. 2012 Nov;13(8):625-37. doi: 10.1007/s10194-012-0477-y. Epub 2012 Aug 31. PMID 22935970
- [Background] Alonso-Blanco C, Fernandez-de-las-Penas C, Morales-Cabezas M, Zarco-Moreno P, Ge HY, Florez-Garcia M. Multiple active myofascial trigger points reproduce the overall spontaneous pain pattern in women with fibromyalgia and are related to widespread mechanical hypersensitivity. Clin J Pain. 2011 Jun;27(5):405-13. doi: 10.1097/AJP.0b013e318210110a. PMID 21368661
- [Derived] Castro-Sanchez AM, Garcia-Lopez H, Fernandez-Sanchez M, Perez-Marmol JM, Leonard G, Gaudreault N, Aguilar-Ferrandiz ME, Mataran-Penarrocha GA. Benefits of dry needling of myofascial trigger points on autonomic function and photoelectric plethysmography in patients with fibromyalgia syndrome. Acupunct Med. 2020 Jun;38(3):140-149. doi: 10.1136/acupmed-2017-011504. Epub 2020 Jan 28. PMID 31986897